CLINICAL TRIAL: NCT02614456
Title: Combination Immunotherapy With Interferon-gamma and Nivolumab for Patients With Advanced Solid Tumors: A Phase 1 Study
Brief Title: Combination of Interferon-gamma and Nivolumab for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Horizon Pharma Ireland, Ltd., Dublin Ireland (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-084
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Interferon-gamma; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interferon-gamma and nivolumab (Experimental): Interferon-gamma (IFN-γ): starting dose 50 mcg/m2 subcutaneously Nivolumab: 3 mg/kg intravenously
  Induction phase: IFN-γ every other day alone for 1 week Combination phase: IFN-γ every other day & Nivolumab every 2 weeks for 3 months Single agent phase: Nivolumab every 3 weeks up to 1 year
  Interventions: Drug: interferon-gamma and nivolumab

INTERVENTIONS:
Drug: interferon-gamma and nivolumab

SUMMARY:
This is a phase I study of combination immunotherapy with IFN-γ and the PD-1 inhibitor nivolumab in patients with advanced solid tumors who have progressed on at least one prior systemic therapy, which may include prior immunotherapy.

DETAILED DESCRIPTION:
This is a phase I study of combination immunotherapy with IFN-γ and the PD-1 inhibitor nivolumab in patients with advanced solid tumors who have progressed on at least one prior systemic therapy, which may include prior immunotherapy. Patients will be treated with a one week induction phase (IP) of IFN-γ, followed by a combination phase (CP) with IFN-γ and nivolumab for three cycles, followed by a single agent phase of only nivolumab for up to one year. The study will primarily assess the safety and tolerability of the combination. Tumor assessments will occur after three cycles of combination therapy, then every three cycles thereafter. Secondary objectives including ORR, PFS, and OS will also be assessed, as will various correlative analyses. Initial accrual will occur using a modified 6+6 design, and if endpoints for safety (using DLT criteria) are met, expansion cohorts in RCC and UC will be opened for up to 15 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologically or cytologically confirmed metastatic solid tumor that has shown clinical or pre-clinical evidence of responding to anti-PD-1 therapy or the capacity to up-regulate PD-L1. These tumor types may include but may not be limited to: RCC, UC, melanoma, non small cell lung cancer (NSCLC), small cell lung cancer, squamous cell cancer of the head and neck (SCCHN), ovarian carcinoma, triple negative breast cancer, gastric cancer, microsatellite instability expressing (MSI-high) colon cancer, hepatocellular carcinoma, mesothelioma, gastrointestinal stromal tumors, endometrial carcinoma, liposarcomas, chondrosarcomas, and uterine sarcomas. Patients with solid tumor types not listed above may be enrolled at the discretion of the Principal Investigator.

   Note: Dose expansion phase will include two cohorts and consist of patients with either metastatic UC or RCC, but must meet all other inclusion criteria.
2. All patients must have received at least one line of systemic therapy in the metastatic setting. Prior immunotherapy is allowed, including prior treatment with nivolumab or another PD-1 inhibitor, as long as the reason for discontinuation of a prior PD-1 inhibitor was not for drug-related toxicity.
3. Patients must have measurable disease per RECIST criteria v. 1.1 as described in detail in section 11.0.
4. Patients must have a site of disease that is amenable to pretreatment and on-treatment core biopies. At least 3 formalin fixed, paraffin embedded (FFPE) slides at five microns each may be collected at each biopsy. Determination of tissue accessibility and quantity will be made by the consenting clinician. Patients must consent to the two study-required biopsy procedures.
5. Age > 18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
7. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count > 1,500/mcL
   * Platelets > 100,000/mcL
   * Total bilirubin < 1.5 times the upper limit of normal (ULN), except patients with Gilbert's syndrome in whom total bilirubin must be <3.0 mg/dL
   * AST/ALT (SGOT/SGPT) < 3 times institutional normal limits
   * Creatinine < 1.5 times the ULN OR Creatinine clearance > 40 mL/min (as measured or calculated by Cockroft-Gault formula)
8. Ability to understand and willingness to sign a written informed consent and HIPAA consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study.
2. Patients may not have any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids or immunosuppressive medications, except for syndromes which would not be expected to recur in the absence of an external trigger. Subjects with vitiligo, type I diabetes mellitus, or residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement are permitted to enroll.
3. Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days prior to first dose of study drug. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease.
4. Patients may not be receiving any other investigational agents.
5. Patients with known active or symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis. Asymptomatic, treated, and/or stable brain metastases, as measured by subsequent radiologic evaluations at least two months apart, are permitted.
6. History of allergic reactions attributed to compound of similar chemical or biologic composition to the agent(s) used in this study.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension or psychiatric illness/social situations that would limit compliance with study requirements.
8. Known human immunodeficiency virus (HIV) positive or history of acquired immune deficiency syndrome (AIDS) or AIDS-defining illness.
9. Known current or a history of hepatitis B or C virus, including chronic and dormant states, unless disease has been treated and confirmed cleared.
10. Any medical condition that in the investigator's opinion could interfere with interpretation of study or toxicity, or increase the risk to the patient related to potential toxicity.
11. Major surgery within 4 weeks of initiation of study drug.
12. Pregnant or breast feeding. Refer to section 4.4 for further detail.
13. A second invasive malignancy requiring active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assesses by CTCAE version 4.03. | 58 weeks
Determine the recommended phase 2 dose (RP2D) based on Dose limiting toxicities | 6 weeks

SECONDARY OUTCOMES:
To evaluate the investigator assessed ORR using standard response evaluation criteria in solid tumors (RECIST) version 1.1 for metastatic renal cell carcinoma. | 2 years
To evaluate the investigator assessed ORR using standard response evaluation criteria in solid tumors (RECIST) version 1.1 for metastatic urothelial cancer. | 2 years
To evaluate median progression free survival (PFS) using Kaplan-Meier curves for metastatic renal cell carcinoma. | 2 years
To evaluate median progression free survival (PFS) using Kaplan-Meier curves for metastatic urothelial cancer. | 2 years
To evaluate median overall survival (OS) using Kaplan-Meier curves for metastatic renal cell carcinoma. | 2 years
To evaluate median overall survival (OS) using Kaplan-Meier curves for metastatic urothelial cancer. | 2 years
To investigate the relationship between PD-L1 expression on tumor cells and on immune cells using IHC and SMI methods. | Baseline
To investigate the relationship between PD-L1 expression on tumor cells and on immune cells using IHC and SMI methods. | week 2
To investigate the relationship between PD-L1 expression on tumor cells and on immune cells using IHC and SMI methods. | week 7

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Zibelman, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Zibelman M, MacFarlane AW 4th, Costello K, McGowan T, O'Neill J, Kokate R, Borghaei H, Denlinger CS, Dotan E, Geynisman DM, Jain A, Martin L, Obeid E, Devarajan K, Ruth K, Alpaugh RK, Dulaimi EA, Cukierman E, Einarson M, Campbell KS, Plimack ER. A phase 1 study of nivolumab in combination with interferon-gamma for patients with advanced solid tumors. Nat Commun. 2023 Jul 27;14(1):4513. doi: 10.1038/s41467-023-40028-z. PMID 37500647